CLINICAL TRIAL: NCT01293084
Title: Acute Inhalation of Hypertonic Saline Does Not Improve Mucociliary Clearance in All Children With Cystic Fibrosis
Brief Title: Hypertonic Saline and Mucociliary Clearance in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Beth L. Laube, Professor, Johns Hopkins University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CFF Account #LAUBE06A0
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Results first posted 2015-09-22 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Cystic Fibrosis
Keywords: mucociliary clearance; children; cystic fibrosis; hypertonic saline
MeSH Terms: conditions — Cystic Fibrosis | interventions — Sodium Chloride; Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 7% saline (Experimental): 5 mL of 7% saline was inhaled once over a 20 minute period.
  Interventions: Drug: 7% saline
- 0.12% saline (Placebo Comparator): 5mL 0.12% saline inhaled once during 20 minutes
  Interventions: Drug: 0.12% saline

INTERVENTIONS:
Drug: 0.12% saline — 5mL of 0.12% saline inhaled once over 20 minutes
  Arms: 0.12% saline
Drug: 7% saline — 5mL 7% saline inhaled once over 20 minutes
  Other Names: hypertonic saline
  Arms: 7% saline

SUMMARY:
Previously, the investigators and others have shown that mucociliary clearance (MCC) is defective in patients with cystic fibrosis (CF) and it is now thought that alterations in airway mucus rheology figure prominently in the impairment. Mucociliary clearance works by trapping toxic particles, bacteria and viruses in the lung mucus and then quickly removing the mucus out of the lungs. Defects in MCC typically lead to the accumulation of mucus in the airways, and this in turn is associated with acute infections, chronic bacterial colonization and chronic inflammation. One treatment strategy that is gaining acceptance as an important therapy for improving MCC in adults with CF is the inhalation of the osmotic stimulus, hypertonic saline (HS). A number of studies have shown that acute inhalation of HS (7% saline) significantly improves MCC in adults with CF and results from a recent study indicate that two weeks of inhaling HS leads to a significant increase in MCC that is sustained for 8 hours post inhalation and is associated with significant improvements in FEV1, FVC and FEF25-75 values. Since MCC in patients with CF appears to be impaired by adulthood, any drug that disrupts or slows the impairment in childhood could prove enormously beneficial in the long-term prognosis of the disease. Nevertheless, no studies have been conducted to determine if HS treatment improves MCC in children with CF. This is most problematic for physicians who care for children with CF who have normal FEV1 and FVC values, since it is unclear if they should treat these children with HS or not. This research study is designed to begin to answer this question. The investigators hypothesize that acute inhalation of hypertonic saline (7%) will improve MCC in CF children with normal pulmonary function. Our hypothesis will be tested in a one-year clinical trial that will be randomized and placebo-controlled. Twelve children with CF who are 7-12 years old and have normal FEV1 and FVC values will participate. Our goal will be to compare MCC in these children on two study visits after acute inhalations of placebo (0.12% saline) or hypertonic saline (HS) (7% saline) aerosol. The investigators predict that MCC values after acute inhalation of 7% HS aerosol will be statistically significantly greater than after placebo inhalation.

DETAILED DESCRIPTION:
Several studies report that mucociliary clearance (MCC) is impaired in adults with CF. Because MCC is an important airway defense mechanism, drugs that slow impairment of MCC in children could prove beneficial in the long-term prognosis of the disease. A few studies have shown that inhalation of hypertonic saline (HS) significantly improves MCC in adults with CF and improvement is associated with increases in pulmonary function and decreases in pulmonary exacerbations. Nevertheless, no studies have examined if HS improves MCC in CF children. This is problematic for physicians who care for CF children with normal pulmonary function, since it is unclear if they should treat with HS or not. This study was designed to begin to answer this question. Twelve children with CF (7-12 yrs; 5 males) and normal pulmonary function (FEV1 and FVC > 90% of predicted values) participated in a screening visit and two study visits. On the screening visit, children underwent an induced sputum test. On the two study visits, they inhaled 0.12% saline (placebo), or HS, in a double-blind, randomized, cross-over study. Following inhalation of placebo or HS, patients inhaled the radioisotope 99mtechnetium and underwent sequential imaging of their lungs with a gamma camera for 90 min and approximately 24 hrs later. Mucociliary clearance was quantified at 60 min (MCC60), 90 min (MCC90) and 24 hrs (MCC24hrs) after inhalation of the radioisotope. Between the 60 min and 90 min measurements, children coughed 30 times.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age 7-12 years old
* Diagnosis of cystic fibrosis by sweat chloride > 60 meq/L, or presence of two CFTR mutations known to cause CF
* Routinely treated with the short-acting bronchodilator albuterol
* FEV1 > 90% of predicted values

Exclusion Criteria:

* FEV1 < 90% of predicted values
* Routine use of hypertonic saline, mannitol, or amiloride
* Allergic bronchopulmonary aspergillosis (ABPA)
* Sputum colonization with Burkholderia cepacia or multiple antibiotic resistant organisms
* Evidence of a pulmonary exacerbation within past two weeks
* Treated with intravenous or oral antibiotics in the past two weeks for a pulmonary exacerbation
* Presence of an acute respiratory illness characterized by:

  * Coughing above baseline values
  * Wheezing
  * Respiratory distress
  * Hemoptysis
* Cannot perform the inhalation maneuvers that are required for drug inhalation or radioaerosol administration

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth L Laube, PhD, Principal Investigator — Johns Hopkins University

REFERENCES:
- [Derived] Laube BL, Sharpless G, Carson KA, Kelly A, Mogayzel PJ Jr. Acute inhalation of hypertonic saline does not improve mucociliary clearance in all children with cystic fibrosis. BMC Pulm Med. 2011 Sep 6;11:45. doi: 10.1186/1471-2466-11-45. PMID 21896198

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data could not be retrieved for the order of randomization.
Groups:
- Children With CF: Children with CF inhaled either 5 mL of 7% saline or 0.12% saline once over 20 minutes. On a second visit, the same children were crossed-over and inhaled either 0.12% saline or 7% saline over 20 minutes. The order of these visits was randomized but the sequence of the randomization is not known.
Period: Overall Study
Arm/Group | Children With CF
Started | 17
Completed | 12
Not Completed | 5
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Children With CF
Number analyzed (Participants) | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 10.5 [8.9 to 12.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 12
FVC (% predicted) [Median (Inter-Quartile Range); unit: percent predicted] | 107 [101.5 to 116.0]
FEV1 (% predicted) [Median (Inter-Quartile Range); unit: percent predicted] | 108 [102.5 to 117.5]
Genotype [Number; unit: participants]
  F508del homozygous | 9
  F508heterozygous | 2
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Mucociliary Clearance at 60 Minutes
Time Frame: 60 minutes
Population: Participants that completed received both 7% saline and 0.12% saline over the duration of the study
Measure: Median (Inter-Quartile Range); unit: percentage mucociliary clearance
Arm/Group | 7% Saline | 0.12% Saline
Number analyzed (Participants) | 12 | 12
percentage mucociliary clearance | 18.6 [12.3 to 27.4] | 15.4 [12.4 to 24.5]
Statistical Analysis 1: Comparison: 7% Saline vs 0.12% Saline; Test type: Superiority or Other; p = 0.62, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 2.2

2. Secondary Outcome: Percent Mucociliary Clearance at 90 Minutes
Time Frame: 90 minutes
Population: Data for participants that completed and received both 7% saline and 0.12% saline.
Measure: Median (Inter-Quartile Range); unit: percentage mucociliary clearance
Arm/Group | 7% Saline | 0.12% Saline
Number analyzed (Participants) | 12 | 12
percentage mucociliary clearance | 27.4 [16.25 to 30.95] | 19.3 [17.3 to 27.8]
Statistical Analysis 1: Comparison: 7% Saline vs 0.12% Saline; Test type: Superiority or Other; p = 0.32, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 2.3

ADVERSE EVENTS:
Arm/Group | 7% Saline | 0.12% Saline
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes